CLINICAL TRIAL: NCT00195247
Title: A Phase 1 Dose Escalation Study of TTI-237 Administered Intravenously Every 3 Weeks in Subjects With Advanced Malignant Solid Tumors
Brief Title: Study Evaluating TTI-237 in Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3162K1-101; NCT00112814 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Neoplasms
Keywords: Tumors; Advanced malignant solid tumors
MeSH Terms: conditions — Neoplasms | interventions — cevipabulin

INTERVENTIONS:
Drug: TTI-237

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and maximum tolerated dose (MTD) of TTI-237 for the treatment of subjects with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of malignant solid tumor with measurable disease
* Life expectancy of at least 12 weeks
* ECOG performance status of 0, 1, or 2

Exclusion Criteria:

* Recent major surgery, radiation therapy or anti-cancer treatment
* History of any other prior malignancy within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-05

PRIMARY OUTCOMES:
Primary purpose is to address the safety and tolerability of TTI-237. Patient will be assessed on an ongoing basis during their participation on the trial.

SECONDARY OUTCOMES:
Preliminary pharmacokinetics (cycle 1 only) and anti-tumor activity of TTI-237 (approximately every 8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - Los Angeles, California
  - Baltimore, Maryland